CLINICAL TRIAL: NCT05749757
Title: The Efficacy and Safety of Acupuncture for Post COVID-19 Fatigue: a Randomized Controlled Trial
Brief Title: Acupuncture for Post COVID-19 Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yuanjie Sun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-013-KY-01
Record Dates: First submitted 2023-02-28; First posted 2023-03-01 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Acupuncture; Post COVID-19 Condition; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Hwato brand disposable acupuncture needles (size 0.30 × 40 mm) and adhesive pads will be used. Acupoints of Guanyuan, Zhongwan, Tianshu, Zusanli, Taixi, Shangyintang, Taiyang, Hegu, Taichong and Shenmen will be selected. Participants will receive a total of 10-session acupuncture treatment during four weeks, three times a week in the first two weeks and twice a week in the last two weeks.
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): Hwato brand disposable placebo needles (with the handle identical to the needles in the acupuncture group and the body at a size 0.30 × 25 mm) and adhesive pads will be used. Acupoints of Guanyuan, Zhongwan, Tianshu, Zusanli, Taixi, Shangyintang, Taiyang, Hegu, Taichong and Shenmen will be selected. Participants will receive a total of 10-session sham acupuncture treatment during four weeks, three times a week in the first two weeks and twice a week in the last two weeks.
  Interventions: Device: Sham Acupuncture

INTERVENTIONS:
Device: Acupuncture — For Shangyitang acupoint, the needle will be inserted towards the direction of nasal tip horizontally to a depth of 10-20mm without any manipulation, and a pad will be adhered afterwards. For other acupoints, the needles will be inserted through adhesive pads to 10-20mm. Needles will be lifted, thrust, and twirled for 3 times to achieve deqi sensation, and will be manipulated every ten minutes during 30-minute maintenance.
  Arms: Acupuncture
Device: Sham Acupuncture — For all the points, the needles will be inserted into adhesive pads without skin penetration. Needles will be lifted, thrust and twirled for 3 times to mimic real acupuncture. No manipulation will be conducted during 30-minute maintenance.
  Arms: Sham Acupuncture

SUMMARY:
The aim of the study is to access the efficacy and safety of acupuncture for post COVID-19 fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75.
* Confirmed COVID-19 infection in the past four weeks to six months, and a negative RT PCR and/or Antigen-Based Rapid Test at present.
* A main complaint of fatigue emerged newly following COVID-19 infection.
* A score of ≥15 on Chalder Fatigue Scale (CFS, score range 0-33).
* Participating the trial volunteerly and providing written informed consent.

Exclusion Criteria:

* Severe anxiety and depression: a score of ≥25 on 17-item Hamilton Rating Scale for Depression (HAMD-17) and/or a score scores >29 on 14-item Hamilton Rating Scale for Anxiety (HAMA-14).
* Significant cognitive dysfunction or suicidal tendency.
* Usage of anti-anxiety and/or anti-depression treatments over the last three months.
* Previously diagnosed hypothyroidism or chronic fatigue syndrome.
* A complication of serious and poorly controlled underlying diseases.
* Having symptoms indicating emergency or severe conditions.
* Concurrent use of other anti-fatigue agents or treatments at present.
* Impaired walking ability.
* Pregnant and/or lactating or planning to get pregnant in the next 4 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the Chalder Fatigue Scale (CFS) score | Week 4
  CFS evaluates physical and mental fatigue with two subscales and 11 items. Total fatigue score is obtained by summing 11 items, which were rated on a four-point Likert scale (0=better than usual, 1=no worse than usual, 2=worse than usual, and 3=much worse than usual). Higher scores indicate more severe fatigue.

SECONDARY OUTCOMES:
The change from baseline in the Chalder Fatigue Scale (CFS) score | Weeks 8, 12, and 16
  CFS evaluates physical and mental fatigue with two subscales and 11 items. Total fatigue score is obtained by summing 11 items, which were rated on a four-point Likert scale (0=better than usual, 1=no worse than usual, 2=worse than usual, and 3=much worse than usual). Higher scores indicate more severe fatigue.
Proportion of participants with a score of less than 15 on CFS | Weeks 4, 8, 12, and 16
  CFS evaluates physical and mental fatigue with two subscales and 11 items. Total fatigue score is obtained by summing 11 items, which were rated on a four-point Likert scale (0=better than usual, 1=no worse than usual, 2=worse than usual, and 3=much worse than usual). Higher scores indicate more severe fatigue.
The change from baseline in the distance of Six-Minute Walk Test (6MWT). | Weeks 4, 8 and 16
  The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface.
The proportion of participants rated as "very much improved" or "much improved" based on the Patient Global Impression-Change (PGI-C). | Weeks 4, 8, 12, and 16
  PGI-C is a 7-point scale, reted by participants themselves, to assess their overall improvement as "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse" or "very much worse".
The change from baseline in the score of physical function dimension of Medical Outcomes Study 36-item Short-Form General Health Survey (SF-36). | Weeks 4, 8, 12, and 16
  Physical functioning of SF-36 is used to assess the health-related quality of life (HRQoL). Physical functioning dimension consists of 10 items with a total score ranging from 0 to 100. Higher scores indicate better HRQoL related to physical functioning.
The change from baseline in the score of Chinese Version of the Work and Social Adjustment Scale (CWSAS). | Weeks 4, 8, 12, and 16
  The CWSAS assesses the impairment of social function in five items of ability to work, home management, social leisure, private leisure, and close relationship. Each item is rated on a 9-point Likert scale from 0 (no impairment) to 8 (very severe impaired). The total score of the scale ranges from 0 to 40, with higher scores indicating more severe psychopathology.
The change from baseline in the score of Montreal Cognitive Assessment (MoCA). | Weeks 4 and 16
  The MoCA is used for rapid assessment of mild cognitive impairment. It consists of 12 subtasks exploring the cognitive domains of memory, visuospatial abilities, executive functions, attention, concentration and working memory, language, temporal and spatial orientation. The total score ranges from 0 (worst performance) to 30 (best performance) and the normal score is no less than 26.
The change from baseline in the score of Patient Health Questionnaire-15 (PHQ-15) score. | Weeks 4 and 16
  PHQ-15 is a self-administered test to assess somatization disorder. It comprises 15 items, and each item scores from 0 ("not bothered at all") to 2 ("bothered a lot").
The change from baseline in the score of Physical Health Questionnaire-9 (PHQ-9) | Weeks 4 and 16
  The PHQ-9 is a nine-item self-rated questionnaire to measure the severity of depressive symptoms over the last two weeks corresponding to the DSM-IV criteria of major depressive disorder. Each item is scored from 0 (not at all) to 3 (nearly every day). Higher scores indicate greater severity of depressive symptoms.
The change from baseline in the score of General Anxiety Disorder-7 (GAD-7). | Weeks 4 and 16
  The GAD-7 is a seven-item self-rated questionnaire to assess the severity of generalized anxiety disorder over the last two weeks according to DSM-IV diagnostic criteria. Each item is rated from 0 (not at all) to 3 (nearly every day). Higher scores indicate greater severity of anxiety symptoms.
The change from baseline in the score of Insomnia Severity Index (ISI). | Weeks 4, 8, 12, and 16
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. A 5-point Likert scale (0-4) is used to rate each item and the total score of ISI ranges from 0 to 28. Higher scores indicate more severe insomnia.

OTHER OUTCOMES:
Expectance assessment | Baseline
  Participants will be asked what do you think the condition of fatigue will be in a month?
Blinding assessment | Within 5 minutes after the either treatment in week 4
  Participants will be asked do you think you have received traditional acupuncture over the past 4 weeks.

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with publication until six months after publication.
  Formal request should be sent to puzhisun@163.com with a methodologically sound proposal. Researchers whose proposal has been approved will sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with publication until until six months after publication.
Access Criteria: Formal request should be sent to puzhisun@163.com with a methodologically sound proposal. Researchers whose proposal has been approved.
  Researchers whose proposal has been approved will sign a data access agreement.